CLINICAL TRIAL: NCT02168231
Title: Abdominal Wall Repair With Strattice in Germany: a Cohort Study (BASE Cohort)
Brief Title: Abdominal Wall Repair With Strattice in Germany: a Cohort Study
Acronym: BASE cohort
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Erasmus Medical Center (Other)
Collaborators: Unfallkrankenhaus Berlin (Other); Johann Wolfgang Goethe University Hospital (Other); Diakoniekrankenhaus Friederikenstift (Other); Krankenhaus Agatharied Hausham (Unknown); Technical University of Munich (Other); St. Josefs-Hospital Wiesbaden GmbH (Other)
Responsible Party: Principal Investigator, Ruth Kaufmann, MD, PhD fellow, Erasmus Medical Center
Other Study IDs: BASE cohort study
Record Dates: First submitted 2014-06-12; First posted 2014-06-20 (Estimated); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Hernia of Abdominal Wall; Biologic Mesh; Strattice
Keywords: Complex abdominal wall hernia; Biologic mesh; Strattice
MeSH Terms: conditions — Hernia, Abdominal | interventions — strattice

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Complex abdominal wall repair Strattice: Complex abdominal wall repair Strattice
  Interventions: Procedure: Complex abdominal wall repair Strattice

INTERVENTIONS:
Procedure: Complex abdominal wall repair Strattice — Not applicable (cross-sectional data from a cohort selected after initial complex abdominal wall surgery with Strattice)
  Other Names: Strattice; Porcine accelular dermal matrix; Non-cross-linked biologic mesh

SUMMARY:
Incisional hernia is the most frequently seen long term complication in surgery causing much morbidity and even mortality in patients. Despite studies on the optimal closing technique for laparotomies, the risk for incisional hernia after midline incision remains about 5-20%. It has been established that implementing a mesh reduces recurrence of the incisional hernia but still the results of repair are often disappointing. Incisional hernias can become increasingly complex due to complicated abdominal wall defects caused by a disturbed anatomy, fistulas, burst abdomen, wound and mesh infections. In these cases it is not save to repair the incisional hernia by means of a synthetic mesh and other augmentation tools need to be implemented.

In the recent years the use of biological meshes has been gaining popularity. Recent reports of the use of collagen-based prosthesis have suggested that they support new vessel growth, do not excite a significant foreign body reaction, form fewer adhesions, are well incorporated into host tissues with minimal wound contraction, and can be used in grossly contaminated wounds with fewer infective complications. Biologic meshes are harvested from a source tissue and processed for medical use but they vary widely in their processing methods. They include tissues of human or animal origins, both chemically cross-linked and non cross-linked processes, and submucosal, pericardial, or dermal tissue sources. Current studies investigating the effectiveness of these meshes are small and have short periods of follow-up. These shortcomings can be explained to high cost of the meshes and unclear indication when to use a biological mesh.

The aim of this study is to investigate the short and long term effects of the Strattice biological mesh. The investigators will also inquire why a biologic mesh was used and what the direct and indirect costs were.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 years or older
* Signed informed consent
* Abdominal wall repair
* Strattice mesh implantation prior to inclusion in BASE cohort

Exclusion Criteria:

* Age under 18 years
* No signed informed consent
* Other operation than abdominal wall repair
* Other mesh than Strattice mesh

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients operated by members of the ROKI group (Arbeitsgruppe für Rekonstruktion komplexer Inzisionaler Hernien); i.e. a group of German hernia surgeons using Strattice for complex abdominal wall surgery. This group of surgeons is willing to share their patient cases with the investigators to achieve more knowledge on this delicate topic.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Incisional hernia recurrence | At one year after initial operation
  This parameter will be assessed by taking a history of the patient, and performing physical examination.
Postoperative complications | Postoperatively, until one year after initial operation
  All postoperative complications and their treatment will be registered.
Survival | Postoperatively; until three years after initial operation
  Any decease postoperatively

SECONDARY OUTCOMES:
EHS incisional hernia classification | Perioperatively (noted just before or just after operation)
  Classification according to Ventral Hernia Working Group classification (Breuing et al. Surgery 2010; 148(3): 544-58).
Mesh explantations | Postoperatively; until three years after initial operation
  Strattice mesh explantation after operation
Additional "abdominal wall repair" operations | Postoperatively; until three years after initial operation
  Additional "abdominal wall (hernia) repair" operations after initial implantation of Strattice
Indication of Strattice usage | Perioperatively (noted just before or just after operation)
  Defined as preoperative conditions that influenced the decision (for instance: presence of stoma, fistulas, abscesses, etc.)
Quality of Life (questionnaire-based) | Postoperatively; measured at one, two and three years after initial operation
  Measured with questionnaires (SF-36, EQ-5D-5L, BIQ)
Health economic analysis | Postoperatively; until one year after initial operation
  Various cost-related parameters
Incisional hernia recurrence | At two and three years after initial operation
  This parameter will be assessed by taking a history of the patient, and performing physical examination.

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Kaufmann, MD, Principal Investigator — Erasmus Medical Center
Locations (6):
- Germany (6):
  - Trauma Hospital Berlin, Berlin
  - Johann Wolfgang Goethe-University, Frankfurt am Main
  - Diakoniekrankenhaus Friederikenstiftung, Hanover
  - Agatharied Hospital, Hausham
  - Klinikum rechts der Isar, Technical University of Munich, München
  - St. Josefs-Hospital Wiesbaden, Wiesbaden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kaufmann R, Isemer FE, Strey CW, Jeekel J, Lange JF, Woeste G. Non-cross-linked biological mesh in complex abdominal wall hernia: a cohort study. Langenbecks Arch Surg. 2020 May;405(3):345-352. doi: 10.1007/s00423-020-01881-4. Epub 2020 Apr 22. PMID 32323007